CLINICAL TRIAL: NCT01672892
Title: A Randomized Phase III Study of Standard vs. IMRT Pelvic Radiation for Post-Operative Treatment of Endometrial and Cervical Cancer (TIME-C)
Brief Title: Standard Versus Intensity-Modulated Pelvic Radiation Therapy in Treating Patients With Endometrial or Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-1203; CDR0000738944; NCI-2012-02001 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-23; First posted 2012-08-27 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Cervical Cancer; Endometrial Cancer; Gastrointestinal Complications; Perioperative/Postoperative Complications; Radiation Toxicity; Urinary Complications; Urinary Tract Toxicity
Keywords: gastrointestinal complications; perioperative/postoperative complications; radiation toxicity; urinary complications; urinary tract toxicity; endometrial clear cell carcinoma; endometrial papillary serous carcinoma; stage IA endometrial carcinoma; stage IB endometrial carcinoma; stage II endometrial carcinoma; stage IIIA endometrial carcinoma; stage IIIB endometrial carcinoma; stage IIIC endometrial carcinoma; endometrial adenocarcinoma; cervical adenocarcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Postoperative Complications; Radiation Injuries | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensity-Modulated Radiation Therapy (Experimental): intensity-modulated radiation therapy (IMRT) to the pelvis of either 45 Gy or 50.4 Gy
  Interventions: Radiation: Standard radiation therapy
- Standard Radiation Therapy (Active Comparator): Standard radiation therapy (4-field) to the pelvis of either 45 Gy or 50.4 Gy
  Interventions: Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: Standard radiation therapy — Patients treated once a day, 5 days a week with a daily fraction size of 1.8 Gy. Whole pelvis treated with a four-field technique (AP/PA/R lateral/L lateral) to 45 or 50.4 Gy at 1.8 Gy/fraction. The dose is prescribed to the isocenter which is defined as the intersection of the four beams and can be normalized to an isodose line between 97-100%. The decision to deliver 45 or 50.4 Gy is at the physician's discretion and must be reported at the time of enrollment.
  Other Names: RT
  Arms: Intensity-Modulated Radiation Therapy
Radiation: intensity-modulated radiation therapy — Patients treated once a day, 5 days a week with a daily fraction size of 1.8 Gy. All targets treated simultaneously. The vaginal planning target volume (PTV) (ITV with 7.0 mm margin) and nodal PTV receives 45 Gy in 25 fractions or 50.4 Gy in 28 fractions. The decision to deliver 45 or 50.4 Gy is at the physician's discretion and must be reported at the time of enrollment.
  Other Names: IMRT
  Arms: Standard Radiation Therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This randomized phase III trial is studying two different methods of radiation and their side effects and comparing how well they work in treating endometrial and cervical cancer after surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if pelvic intensity-modulated radiation therapy (IMRT) reduces acute gastrointestinal toxicity in the 5th week (after 23-25 fractions) of pelvic radiation as measured with the expanded prostate cancer index composite (EPIC) instrument.

Secondary

* To determine if grade 2+ gastrointestinal toxicity (Common Terminology Criteria for Adverse Events version 4.0 [CTCAE v. 4.0]) is reduced with IMRT compared to conventional whole-pelvis radiation therapy (WPRT).
* To determine if grade 2+ hematologic toxicity (CTCAE v. 4.0) is reduced with IMRT compared to conventional WPRT.
* To determine if urinary toxicity is reduced with IMRT using the EPIC urinary domain.
* To validate EPIC bowel and urinary domains in women undergoing either IMRT pelvic radiation treatment or four-field pelvic radiation treatment for endometrial or cervical cancer.
* To assess the impact of pelvic IMRT on quality of life using the Functional Assessment of Cancer Therapy-General (FACT-G) with cervix subscale.
* To determine if there is any difference in local-regional control, disease-free survival, and overall survival between patients treated with IMRT as compared to conventional WPRT.
* To perform a health-utilities analysis to measure the financial impact of pelvic IMRT via the EQ-5D instrument.
* To identify molecular predictors of radiation toxicity and novel circulating cancer biomarkers.

OUTLINE: This is a multicenter study. Patients are stratified according to type of cancer (endometrial vs cervical), chemotherapy (none vs 5 courses of weekly cisplatin at 40 mg/m²), and radiation dose (45 Gy vs 50.4 Gy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard (3-dimensional) radiation therapy 5 days a week for up to 5-6 weeks.
* Arm II: Patients undergo intensity-modulated radiation therapy (IMRT) 5 days a week for up to 5-6 weeks.

Some patients receive cisplatin IV over 1 hour on day 1. Treatment continues weekly for 5 weeks, concurrently with radiation therapy, in the absence of unacceptable toxicity or disease progression.

Tissue and blood samples may be collected for biomarker and correlative analysis.

Quality of life may be assessed by questionnaires (including the Expanded Prostate Cancer Index Composite [EPIC], the Functional Assessment of Cancer Therapy-General [FACT-G, Version 4], the EQ-5D, and the Common Toxicity Criteria Adverse Events - Patient-Reported Outcome [PRO-CTCAE]) instruments at baseline and periodically during and after study therapy.

After completion of study therapy, patients are followed every 6 months for the first 2 years and then annually for 5 years.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically proven diagnosis of endometrial or cervical cancer.
2. Patients must have undergone a hysterectomy (total abdominal hysterectomy, vaginal hysterectomy or radical hysterectomy or total laparoscopic hysterectomy) for carcinoma of the cervix or endometrium within 49 days prior to registration. Performance of a bilateral salpingooophorectomy will be at the treating surgeon's discretion.
3. Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

   * 3.1 History/physical examination within 45 days prior to registration;
   * 3.2 CT, MRI or positron emission tomography - computed tomography (PET-CT) including the abdomen and pelvis should be performed for initial radiological staging. This may be performed pre- or post-surgery within 90 days prior to registration. Imaging performed post-operatively should show no evidence of residual disease. Any evidence of malignancy identified on pre-operative imaging should have been completely resected surgically prior to protocol treatment.
   * 3.3 Chest CT or chest x-ray must be performed within 90 days prior to registration (unless a PET-CT has been performed)
4. Zubrod Performance Status 0-2
5. Age ≥ 18;
6. Complete blood count (CBC)/differential obtained within 14 days prior to registration on study, with adequate bone marrow function defined as follows:

   * 6.1 Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
   * 6.2 Platelets ≥ 100,000 cells/mm3;
   * 6.3 Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
7. For patients receiving chemotherapy:

7.1 Within 14 days prior to registration, serum creatinine ≤ 1.5 mg/dL and calculated creatinine clearance ≥ 50 cc/min. Both tests must be within these limits. The creatinine clearance should be calculated using the Cockcroft-Gault formula: (See Section 7.3.1) 7.2 Aspartate aminotransferase (AST) ≤ 2 x upper limit of normal (ULN) 7.3 Bilirubin ≤ 2 x ULN 7.4 Alkaline phosphatase, Mg, blood urea nitrogen (BUN) and electrolytes must be obtained and recorded 8 Endometrial Cancer: 8.1 Patients with the following histologic features are eligible for pelvic radiation therapy without weekly cisplatin:

* <50% myometrial invasion, grade 3 adenocarcinoma without uterine serous carcinoma (USC) or clear cell histology
* ≥50% myometrial invasion grade 1-2 adenocarcinoma without USC or clear cell histology 8.2 Patients with the following histologic features may be treated with pelvic radiation with or without weekly cisplatin. The decision to add weekly cisplatin for these patients is at the treating physician's discretion:
* ≥50% myometrial invasion, grade 3 including USC and clear cell carcinoma.
* International Federation of Gynecology and Obstetrics (FIGO) 2009 stage II endometrial cancer of any grade including USC and clear cell carcinoma.
* FIGO 2009 IIIC1 (pelvic lymph node positive only, para-aortic nodes negative if removed) including USC and clear cell carcinoma. Note: If para-aortic nodes are not removed, CT abdomen or PET CT must demonstrate no evidence of lymphadenopathy. 9. Cervical Cancer: 9.1 Patients with the following pathology findings may be treated with pelvic radiation with or without weekly cisplatin at the treating physician's discretion. The decision to add weekly cisplatin for these patients is at the treating physician's discretion. 9.1.1 Patients with intermediate risk features including two of the following histologic findings after radical hysterectomy:
* 1/3 or more stromal invasion
* Lymph-vascular space invasion
* Large clinical tumor diameter (> 4 cm) 9.1.2 Patients with cervical cancer treated with a simple hysterectomy with negative margins 9.2 Patients with any of the following criteria following radical hysterectomy are eligible for this study and must receive weekly cisplatin:
* Positive resected pelvic nodes and para-aortic nodes negative if removed. Note: If para-aortic nodes are not removed, CT abdomen or PET CT must demonstrate no evidence of lymphadenopathy.
* Microscopic parametrial invasion with negative margins. 10. Patient must provide study specific informed consent prior to study entry. 11. Willingness and ability to complete the bowel and urinary domains of the EPIC prior to registration

Exclusion criteria:

1. Patients with para-aortic nodal disease or who require extended field radiotherapy beyond the pelvis.
2. Patients with histology consisting of endometrial stromal sarcoma, leiomyosarcoma or malignant mixed mullerian mixed tumor (MMMT or carcinosarcoma)
3. Patients who exceed the weight/size limits of the treatment table or CT scanner.
4. Mental status changes or bladder control problems that make the patient unable to comply with bladder-filling instructions.
5. Patients with evidence of metastatic disease outside of the pelvis.
6. Patients with positive or close (< 3 mm) resection margins
7. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years.
8. Prior radiation therapy to the pelvis
9. Patients with active inflammatory bowel disease. 10 Severe, active co-morbidity, defined as follows:

   * 10.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   * 10.2 Transmural myocardial infarction within the last 6 months
   * 10.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * 10.4 Other major medical illness which requires hospitalization or precludes study therapy at the time of registration
   * 10.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however,that laboratory test coagulation parameters are not required for entry into this protocol
   * 10.6 Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immunocompromised patients.

11. Patients with prior treatment with platinum-based chemotherapy 12. Women who are breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Klopp, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (137):
- United States (129):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - California Cancer Center - North Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Feather River Cancer Center, Paradise, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - University of California at Davis Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Leeward Radiation Oncology Center, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Franciscan Saint Margaret Health-Dyer Campus, Dyer, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Franciscan Saint Margaret Health-Hammond Campus, Hammond, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - The Nebraska Medical Center, Omaha, Nebraska
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - South Atlantic Radiation Oncology, Supply, North Carolina
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Saint Francis Hospital, Federal Way, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (6):
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Yeung AR, Pugh SL, Klopp AH, Gil KM, Wenzel L, Westin SN, Gaffney DK, Small W Jr, Thompson S, Doncals DE, Cantuaria GHC, Yaremko BP, Chang A, Kundapur V, Mohan DS, Haas ML, Kim YB, Ferguson CL, Deshmukh S, Bruner DW, Kachnic LA. Improvement in Patient-Reported Outcomes With Intensity-Modulated Radiotherapy (RT) Compared With Standard RT: A Report From the NRG Oncology RTOG 1203 Study. J Clin Oncol. 2020 May 20;38(15):1685-1692. doi: 10.1200/JCO.19.02381. Epub 2020 Feb 19. PMID 32073955
- [Result] Gil KM, Pugh SL, Klopp AH, Yeung AR, Wenzel L, Westin SN, Gaffney DK, Small W Jr, Thompson S, Doncals DE, Cantuaria GHC, Yaremko BP, Chang A, Kundapur V, Mohan DS, Haas ML, Kim YB, Ferguson CL, Deshmukh S, Kachnic LA, Bruner DW. Expanded validation of the EPIC bowel and urinary domains for use in women with gynecologic cancer undergoing postoperative radiotherapy. Gynecol Oncol. 2019 Jul;154(1):183-188. doi: 10.1016/j.ygyno.2019.04.682. Epub 2019 May 16. PMID 31104905
- [Result] Klopp AH, Yeung AR, Deshmukh S, Gil KM, Wenzel L, Westin SN, Gifford K, Gaffney DK, Small W Jr, Thompson S, Doncals DE, Cantuaria GHC, Yaremko BP, Chang A, Kundapur V, Mohan DS, Haas ML, Kim YB, Ferguson CL, Pugh SL, Kachnic LA, Bruner DW. Patient-Reported Toxicity During Pelvic Intensity-Modulated Radiation Therapy: NRG Oncology-RTOG 1203. J Clin Oncol. 2018 Aug 20;36(24):2538-2544. doi: 10.1200/JCO.2017.77.4273. Epub 2018 Jul 10. PMID 29989857
- [Derived] Yeung AR, Deshmukh S, Klopp AH, Gil KM, Wenzel L, Westin SN, Konski AA, Gaffney DK, Small W Jr, Thompson JS, Doncals DE, Cantuaria GHC, D'Souza DP, Chang A, Kundapur V, Mohan DS, Haas ML, Kim YB, Ferguson CL, Pugh SL, Kachnic LA, Bruner DW. Intensity-Modulated Radiation Therapy Reduces Patient-Reported Chronic Toxicity Compared With Conventional Pelvic Radiation Therapy: Updated Results of a Phase III Trial. J Clin Oncol. 2022 Sep 20;40(27):3115-3119. doi: 10.1200/JCO.21.02831. Epub 2022 Aug 12. PMID 35960897
- Available data/document: Individual Participant Data Set: NCT01672892-D1 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Started | 137 | 152
Eligible Population | 130 | 149
Adverse Event Population (Eligible participants with adverse event data collected anytime during the study.) | 125 | 144
Completed (Participants contributing data to any results are considered to have completed the study.) | 130 | 149
Not Completed | 7 | 3
Not completed — Protocol Violation | 7 | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy | Total
Number analyzed (Participants) | 129 | 149 | 278
Age, Continuous [Median (Full Range); unit: years] | 62 [28 to 82] | 61 [29 to 83] | 61 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 149 | 278
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Acute Gastrointestinal Toxicity, as Measured by Change in Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain Score at 5 Weeks From the Start of Pelvic Radiation
Description: The primary endpoint is change in acute GI toxicity, as measured by the EPIC bowel domain, from baseline to 5 weeks after the first fraction of radiation is delivered. The EPIC has four domains (bowel, urinary, sexual, and hormonal) that have been validated separately, which allows use of only the domains of interest. The EPIC bowel domain consists of 14 items and has a function subscale (7 items) and bother subscale (7 items). For each domain, responses form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, where higher scores correspond to better quality of life. At least 80% of the items in a domain or subscale of the domain must be completed in order to compute the score. Change was calculated as follow-up score - baseline score so a negative change score indicates a decline in function.
Time Frame: Baseline and week 5 of RT
Population: Questionnaires were not completed by all eligible participants. Therefore, only 107/130 had data at both baseline and week 5 on the Intensity-Modulated Radiation Therapy arm, and only 126/149 had data at both baseline and week 5 on the Standard Radiation Therapy arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 107 | 126
units on a scale | -18.6 (18.7) | -23.6 (19.4)
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Since there is no prior data using this tool in this patient population, an effect size of 0.4 was chosen to calculate sample size. Based on a two-sample t-test with one interim look and a two-sided alpha=0.05, a sample size of 225 is needed to achieve 85% statistical power. Assuming an attrition rate of 10% and noncompliance of 10%, 281 patients were required in order to ensure 225 evaluable patients for the primary endpoint analysis; Test type: Superiority; p = 0.0476, t-test, 1 sided

2. Secondary Outcome: Percentage of Patients With Acute Grade 2+ GI Toxicity at 5 Weeks From the Start of Treatment
Description: Adverse events are graded using CTCAE v4.0. Grade refers to the severity of the AE. The Common Terminology Criteria for Adverse Events (CTCAE) v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: Baseline to Week 5 of RT
Population: Adverse event data was not obtained from all eligible participants at 5 weeks from treatment start. Therefore, only 122/130 had data on the Intensity-Modulated Radiation Therapy arm, and only 136/149 had data at on the Standard Radiation Therapy arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 122 | 136
percentage of participants | 26.2 [18.4 to 34.4] | 22.1 [15.1 to 29.0]
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Test type: Superiority; p = 0.4338, Binomial test of proportions; 2-sided significance level = 0.05

3. Secondary Outcome: Urinary Toxicity, as Measured by Change in EPIC Urinary Domain
Description: The primary endpoint is change in acute GI toxicity, as measured by the EPIC urinary domain, from baseline to 5 weeks after the first fraction of radiation is delivered. The EPIC has four domains (bowel, urinary, sexual, and hormonal) that have been validated separately, which allows use of only the domains of interest. The EPIC urinary domain consists of 12 items and has a function subscale (5 items) and bother subscale (7 items). For each domain, responses form a Likert scale and multi-item scale scores are transformed linearly to a 0-100 scale, where higher scores correspond to better quality of life. At least 80% of the items in a domain or subscale of the domain must be completed in order to compute the score. Change was calculated as follow-up score - baseline score so a negative change score indicates a decline in function.
Time Frame: Baseline, week 3 and 5 of RT, and 4-6 weeks after RT
Population: Questionnaires were not completed by all eligible participants. Therefore, data was only collected from: Arm A- 110/130 at baseline and week 3, 107/130 at baseline and week 5, 99/130 at baseline and 4-6 weeks; Arm B- 127/149 at baseline and week 3, 126/149 at baseline and week 5, 121/149 at baseline and 4-6 week.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intensity-Modulated Radiation Therapy (A): Intensity-modulated radiation therapy (IMRT) to the pelvis of either 45 Gy or 50.4 Gy
- Standard Radiation Therapy (B): Standard radiation therapy (4-field) to the pelvis of either 45 Gy or 50.4 Gy
Arm/Group | Intensity-Modulated Radiation Therapy (A) | Standard Radiation Therapy (B)
Number analyzed (Participants) | 130 | 149
score on a scale
  Week 3 of RT: number analyzed (Participants) | 110 | 127
  Week 3 of RT | -2.5 (11.3) | -6.0 (14.5)
  Week 5 of RT: number analyzed (Participants) | 107 | 126
  Week 5 of RT | -5.6 (15.3) | -10.4 (17.5)
  4-6 Weeks Post-RT: number analyzed (Participants) | 99 | 121
  4-6 Weeks Post-RT | -2.7 (13.0) | -4.1 (12.1)
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy (A) vs Standard Radiation Therapy (B); Week 3 of RT; Test type: Superiority; p = 0.04, t-test, 2 sided; 2-sided significance level of 0.05
Statistical Analysis 2: Comparison: Intensity-Modulated Radiation Therapy (A) vs Standard Radiation Therapy (B); Week 5 of RT; Test type: Superiority; p = 0.03, t-test, 2 sided; 2-sided significance level of 0.05
Statistical Analysis 3: Comparison: Intensity-Modulated Radiation Therapy (A) vs Standard Radiation Therapy (B); 4-6 weeks post-RT; Test type: Superiority; p = 0.41, t-test, 2 sided; 2-sided significance level of 0.05

4. Secondary Outcome: Quality of Life, as Measured by Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G) and FACT-Cx (Cervix) Subscale
Description: The FACT-G is a validated, 27-item measure where a higher score represents higher QOL. In addition to a total QOL score, subscale scores for physical, functional, social and emotional well-being are produced. There are 5 responses options, with 0=Not a lot and 4=Very much. All items in a subscale are added together to obtain subscale totals. Scores range from 0-108 for the FACT-G total score, 0-28 for physical, social, functional, and 0-24 for emotional subscale. Certain items must be reversed before it is added by subtracting the response from 4. Subscale totals are summed to form the FACT-G total score. The FACT-Cx is 5-items, with score ranging 0-60, but is not included in total FACT-G. Each subscale requires >= 50% of items completed and overall response rate must be greater than 80%. If items are missing, the subscale scores can be prorated. Change calculated as follow-up score - baseline score so that a negative change score indicates a decline in function.
Time Frame: Before study start, Week 5 of RT, 4-6 Weeks after RT, 1 year from start of RT and 3 years from start of RT
Population: Questionnaires were not completed by all eligible participants. Therefore, the number of participants reported below are the number with the relevant questions answered at baseline and the given time point on each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 130 | 149
score on a scale
  FACT-G total - 5 weeks: number analyzed (Participants) | 85 | 104
  FACT-G total - 5 weeks | -6.4 (12.7) | -7.6 (13.4)
  FACT-G total 4-6 weeks post-RT: number analyzed (Participants) | 80 | 100
  FACT-G total 4-6 weeks post-RT | -0.2 (11.7) | 0.5 (13.9)
  FACT-Cx subscale - 5 weeks: number analyzed (Participants) | 87 | 104
  FACT-Cx subscale - 5 weeks | -2.7 (6.1) | -4.9 (6.5)
  FACT-Cx subscale - 4-6 weeks post-RT: number analyzed (Participants) | 81 | 100
  FACT-Cx subscale - 4-6 weeks post-RT | -0.3 (5.7) | 0.4 (5.7)
  Physical subscale - 5 weeks: number analyzed (Participants) | 86 | 106
  Physical subscale - 5 weeks | -4.2 (6.0) | -6.1 (6.1)
  Physical - subscale - 4-6 weeks post-RT: number analyzed (Participants) | 81 | 101
  Physical - subscale - 4-6 weeks post-RT | -1.1 (4.9) | -1.2 (4.8)
  Functional subscale - 5 weeks: number analyzed (Participants) | 87 | 105
  Functional subscale - 5 weeks | -2.1 (5.7) | -1.6 (5.9)
  Functional - subscale - 4-6 weeks post-RT: number analyzed (Participants) | 81 | 100
  Functional - subscale - 4-6 weeks post-RT | -0.1 (5.0) | 0.6 (5.4)
  Emotional subscale - 5 weeks: number analyzed (Participants) | 87 | 106
  Emotional subscale - 5 weeks | 0.7 (3.5) | 0.9 (3.7)
  Emotional subscale - 4-6 weeks post-RT: number analyzed (Participants) | 81 | 101
  Emotional subscale - 4-6 weeks post-RT | 1.1 (3.1) | 1.9 (3.7)
  Social subscale - 5 weeks: number analyzed (Participants) | 85 | 106
  Social subscale - 5 weeks | -0.9 (5.4) | -0.6 (5.2)
  Social subscale - 4-6 weeks post-RT: number analyzed (Participants) | 80 | 101
  Social subscale - 4-6 weeks post-RT | 0.0 (4.8) | -0.8 (6.4)
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; FACT-G total score - 5 weeks; Test type: Superiority; p = 0.54, t-test, 2 sided; 2-sided significance level = 0.05
Statistical Analysis 2: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; FACT-G total score - 4-6 weeks post RT; Test type: Superiority; p = 0.72, t-test, 2 sided; FACT-G total score - 4-6 weeks post RT
Statistical Analysis 3: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; FACT-Cx subscale score - 5 weeks; Test type: Superiority; p = 0.01, t-test, 2 sided; 2-sided significance level = 0.05
Statistical Analysis 4: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; FACT-Cx subscale score - 4-6 weeks post RT; Test type: Superiority; p = 0.45, t-test, 2 sided; 2-sided significance level = 0.05
Statistical Analysis 5: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Physical subscale score - 5 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 6: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Physical subscale score - 4-6 weeks post RT; Test type: Superiority; p = 0.9, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 7: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Functional subscale score - 5 weeks; Test type: Superiority; p = 0.55, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 8: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Functional subscale score - 4-6 weeks post RT; Test type: Superiority; p = 0.35, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 9: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Emotional subscale score - 5 weeks; Test type: Superiority; p = 0.66, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 10: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Emotional subscale score - 4-6 weeks post RT; Test type: Superiority; p = 0.09, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 11: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Social subscale score - 5 weeks; Test type: Superiority; p = 0.66, t-test, 2 sided; 2-sided significance level = 0.0125
Statistical Analysis 12: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Social subscale score - 4-6 weeks post RT; Test type: Superiority; p = 0.35, t-test, 2 sided; 2-sided significance level = 0.0125

5. Secondary Outcome: Health Utilities, as Measured by Change From Baseline in EQ-5D
Description: The EQ-5D is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). Health states are defined by the combination of the leveled responses to the 5 dimensions, generating 243 health states to which unconsciousness and death are added. The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm 10-point interval scale. Worst imaginable health state is scored as 0 at the bottom of the scale, and best imaginable health state is scored as 100 at the top. Both the 5-item index score and the VAS score are transformed into a utility score between 0 (worst health state) and 1 (best health state). Change from baseline is calculated as score at the timepoint of interested - baseline score.
Time Frame: Baseline, week 5 of RT, 4-6 weeks after RT
Population: Questionnaires were not completed by all eligible participants. Therefore, data was only collected from: Intensity-Modulated Radiation Therapy arm: 78/130 at baseline and week 5, 74/130 at baseline and 4-6 weeks post-RT; Standard Radiation Therapy arm: 91/149 at baseline and week 5, 89/149 at baseline and 4-6 weeks post-RT.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 130 | 149
score on a scale
  5 weeks: number analyzed (Participants) | 78 | 91
  5 weeks | 0 (0.2) | 0 (0.2)
  4-6 weeks post-RT: number analyzed (Participants) | 74 | 89
  4-6 weeks post-RT | 0 (0.1) | 0 (0.1)
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; 5 weeks; Test type: Superiority; p = 0.61, t-test, 2 sided; 2-sided significance level = 0.05
Statistical Analysis 2: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; 4-6 weeks post-RT; Test type: Superiority; p = 0.67, t-test, 2 sided; 2-sided significance level = 0.05

6. Secondary Outcome: Local-regional Recurrence
Description: Local recurrence is defined as a disease in the radiation treatment field. This can include a local vaginal recurrence or nodal disease within the field. Para-aortic recurrence is defined as new lymphadenopathy in the para-aortic distribution. Local-regional control time is defined as time from randomization to the date of local recurrence, last known follow-up (censored), or death (competing risk). Local-regional recurrence rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year rates are provided. Analysis occurred after all patients had been on study for at least 3 years.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 37.8 months.
Population: Eligible participants [later analysis]
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 130 | 149
percentage of participants | 3.5 [1.1 to 8.1] | 2.2 [0.6 to 5.7]
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Test type: Superiority; p = 0.81, Gray's test; Two-sided significance level = 0.05

7. Secondary Outcome: Disease-free Survival
Description: Disease (progression) is defined as local recurrence, para-aortic recurrence, or distant metastasis. Local recurrence is defined as a disease in the radiation treatment field. Para-aortic recurrence is defined as new lymphadenopathy in the para-aortic distribution. Distant metastasis is defined as involvement of another organ or peritoneal disease. Disease-free survival time is defined as time from randomization to the date of progression, death, or last known follow-up (censored). Disease-free survival rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year rates are provided. Analysis occurred after all patients had been on study for at least 3 years.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 37.8 months.
Population: Eligible participants [later analysis]
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 130 | 149
percentage of participants | 85.5 [79.2 to 91.9] | 80.8 [74.2 to 87.3]
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Test type: Superiority; p = 0.21, Log Rank; Two-side significance level = 0.05; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.82 to 2.35] — Reference level = Intensity-Modulated Radiation Therapy

8. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause or last known follow-up (censored). Survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Three-year rates are provided. Analysis occurred after all patients had been on study for at least 3 years.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 37.8 months.
Population: Eligible participants [later analysis]
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 130 | 149
percentage of participants | 92.4 [87.7 to 97.2] | 97.0 [94.1 to 99.9]
Statistical Analysis 1: Comparison: Intensity-Modulated Radiation Therapy vs Standard Radiation Therapy; Test type: Superiority; p = 0.53, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.32 to 1.79] — Reference level = Intensity-Modulated Radiation Therapy

9. Secondary Outcome: Identification of Molecular Predictors of Radiation Toxicity and Novel Circulating Cancer Biomarkers
Time Frame: Outcome measure will not be analyzed
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Standardized Cronbach's Alpha for EPIC Bowel and Urinary Domains (Validation - Internal Consistency Reliability)
Description: The EPIC bowel domain consists of 14 items and has a function subscale (7 items) and bother subscale (7 items). The EPIC urinary domain consists of 12 total items and 4 subscales, functional (5 items), bother (7), incontinence (4) and irritative/obstructive (7). For each item, responses form a Likert scale which are transformed to a 0-100 scale in which higher scores correspond to better quality of life. A domain score is the average of the transformed item scores. At least 80% of the items in a domain or subscale of the domain must be completed in order to compute the score. Cronbach's alpha is an internal consistency estimate of reliability of psychometric test scores and is a function of the number of items in a test, the average covariance between item-pairs, and the variance of the total score. An alpha of 0.60-0.79 was to be considered acceptable reliability; higher than 0.8 was to be considered good reliability.
Time Frame: Baseline and week 5 of RT
Population: Questionnaires were not completed by all eligible participants. Therefore, for both domains data was only collected from: 277/279 (arms combined) at baseline, 241/279 at week 5. [later analysis]
Measure: Number; unit: standard deviation
Groups:
- All Participants: Participants from both treatment arms combined.
Arm/Group | All Participants
Number analyzed (Participants) | 279
standard deviation
  Bowel Domain Baseline: number analyzed (Participants) | 277
  Bowel Domain Baseline | 0.77
  Bowel Domain Week 5: number analyzed (Participants) | 241
  Bowel Domain Week 5 | 0.89
  Urinary Domain Baseline: number analyzed (Participants) | 277
  Urinary Domain Baseline | 0.84
  Urinary Domain Week 5: number analyzed (Participants) | 241
  Urinary Domain Week 5 | 0.89

11. Secondary Outcome: Spearman's Correlation Coefficient for EPIC Bowel Domain vs. Urinary Domains (Validation - Conceptual Independence)
Description: The EPIC bowel domain consists of 14 items and has a function subscale (7 items) and bother subscale (7 items). The EPIC urinary domain consists of 12 total items and 4 subscales, functional (5 items), bother (7), incontinence (4) and irritative/obstructive (7). For each item, responses form a Likert scale which are transformed to a 0-100 scale in which higher scores correspond to better quality of life. A domain score is the average of the transformed item scores. At least 80% of the items in a domain or subscale of the domain must be completed in order to compute the score. Spearman's rank correlation coefficient is a nonparametric measure of rank correlation between two variables with a value between +1 and -1, where 1 is total positive rank correlation, 0 is no rank correlation, and -1 is total negative rank correlation.
Time Frame: Baseline and week 5 of RT
Population: as for outcome 10
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 279
correlation coefficient
  Baseline: number analyzed (Participants) | 277
  Baseline | 0.41
  Week 5: number analyzed (Participants) | 241
  Week 5 | 0.45
Statistical Analysis 1: Comparison: All Participants; Baseline; Test type: Other; p < 0.0001, nonparametric one-sample t-test
Statistical Analysis 2: Comparison: All Participants; Week 5; Test type: Other; p < 0.0001, nonparametric one-sample t-test

12. Secondary Outcome: Pearson Correlation Coefficient for EPIC Bowel and Urinary Domains vs. FACT-G Total Score (Validation - Criterion Validity)
Description: The EPIC bowel domain and urinary domains consist of 14 and 12 items, respectively. For each item, responses form a Likert scale which are transformed to a 0-100 scale in which higher scores correspond to better quality of life (QOL). A domain score is the average of the transformed item scores. At least 80% of the items in a domain must be completed in order to compute the score. The FACT-G is 27-item measure. Higher scores represent higher QOL. Each item has 5 responses options, 0=Not a lot and 4=Very much. Items are added together for the total score, ranging from 0-108. Certain items must be reversed before adding by subtracting the response from 4. The Pearson correlation coefficient is a measure of the linear correlation between two variables with a value between +1 and -1, where 1 is total positive linear correlation, 0 is no linear correlation, and -1 is total negative linear correlation.
Time Frame: Baseline and week 5 of RT
Population: Participants with baseline EPIC and FACT-G scores [later analysis] Questionnaires were not completed by all eligible participants. Therefore, for both domains only 231/279 (arms combined) participants had both FACT-G and EPIC data at baseline, and 199/279 participants had both FACT-G and EPIC data at week 5. [later analysis]
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 279
correlation coefficient
  Bowel Baseline: number analyzed (Participants) | 231
  Bowel Baseline | 0.44
  Bowel Week 5: number analyzed (Participants) | 199
  Bowel Week 5 | 0.44
  Urinary Baseline: number analyzed (Participants) | 231
  Urinary Baseline | 0.39
  Urinary Week 5: number analyzed (Participants) | 199
  Urinary Week 5 | 0.43
Statistical Analysis 1: Comparison: All Participants; Bowel domain at baseline; Test type: Other; p < 0.0001, One-sample t-test
Statistical Analysis 2: Comparison: All Participants; Bowel domain at week 5; Test type: Other; p < 0.0001, One-sample t-test
Statistical Analysis 3: Comparison: All Participants; Urinary domain at baseline; Test type: Other; p < 0.0001, One-sample t-test
Statistical Analysis 4: Comparison: All Participants; Urinary domain at week 5; Test type: Other; p < 0.0001, One-sample t-test

13. Secondary Outcome: Mean Change From Baseline in EPIC Bowel and Urinary Domain (Validation - Sensitivity to Treatment)
Description: The EPIC bowel domain and urinary domains consist of 14 and 12 items, respectively. For each item, responses form a Likert scale which are transformed to a 0-100 scale in which higher scores correspond to better quality of life (QOL). A domain score is the average of the transformed item scores. At least 80% of the items in a domain must be completed in order to compute the score. Difference is calculated as baseline - week 5.
  A positive change score represents a decline in function.
Time Frame: Baseline and week 5 of RT
Population: Questionnaires were not completed by all eligible participants. Therefore, for both domains only 234/279 (arms combined) participants had data at both baseline and week 5. [later analysis]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 279
score on a scale
  Bowel Domain: number analyzed (Participants) | 234
  Bowel Domain | 21.37 (19.11)
  Urinary Domain: number analyzed (Participants) | 234
  Urinary Domain | 8.11 (16.98)
Statistical Analysis 1: Comparison: All Participants; Bowel domain; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: All Participants; Urinary domain; Test type: Other; p < 0.0001, Paired t-test

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 37.8 months. [Later analysis]
Description: Eligible participants with adverse event data. (With the longer follow-up, adverse event data was collected from more participants compared to outcome measure 2. )
Arm/Group | Intensity-Modulated Radiation Therapy | Standard Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 1/125 | 2/144
Other Adverse Events (participants affected / at risk) | 122/125 | 136/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensity-Modulated Radiation Therapy (N=125) | Standard Radiation Therapy (N=144)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensity-Modulated Radiation Therapy (N=125) | Standard Radiation Therapy (N=144)
Anemia (Blood and lymphatic system disorders) | 26 | 17
Tinnitus (Ear and labyrinth disorders) | 7 | 15
Blurred vision (Eye disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 46 | 57
Bloating (Gastrointestinal disorders) | 12 | 13
Constipation (Gastrointestinal disorders) | 26 | 26
Diarrhea (Gastrointestinal disorders) | 96 | 113
Dyspepsia (Gastrointestinal disorders) | 8 | 8
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 10 | 10
Nausea (Gastrointestinal disorders) | 49 | 62
Proctitis (Gastrointestinal disorders) | 10 | 9
Rectal hemorrhage (Gastrointestinal disorders) | 5 | 10
Rectal pain (Gastrointestinal disorders) | 11 | 13
Vomiting (Gastrointestinal disorders) | 16 | 28
Edema limbs (General disorders) | 20 | 17
Fatigue (General disorders) | 91 | 94
Pain (General disorders) | 20 | 20
Urinary tract infection (Infections and infestations) | 13 | 10
Dermatitis radiation (Injury, poisoning and procedural complications) | 8 | 16
Lymphocyte count decreased (Investigations) | 14 | 17
Neutrophil count decreased (Investigations) | 8 | 8
Platelet count decreased (Investigations) | 11 | 6
Weight loss (Investigations) | 10 | 9
White blood cell decreased (Investigations) | 21 | 16
Anorexia (Metabolism and nutrition disorders) | 26 | 27
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 1
Hypokalemia (Metabolism and nutrition disorders) | 7 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 5
Hyponatremia (Metabolism and nutrition disorders) | 10 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 14
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 8
Headache (Nervous system disorders) | 16 | 14
Paresthesia (Nervous system disorders) | 15 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 13
Anxiety (Psychiatric disorders) | 10 | 12
Depression (Psychiatric disorders) | 9 | 12
Insomnia (Psychiatric disorders) | 12 | 19
Cystitis noninfective (Renal and urinary disorders) | 9 | 10
Renal and urinary disorders - Other (Renal and urinary disorders) | 10 | 8
Urinary frequency (Renal and urinary disorders) | 37 | 48
Urinary incontinence (Renal and urinary disorders) | 23 | 21
Urinary tract pain (Renal and urinary disorders) | 12 | 22
Urinary urgency (Renal and urinary disorders) | 13 | 24
Pelvic pain (Reproductive system and breast disorders) | 22 | 30
Vaginal discharge (Reproductive system and breast disorders) | 7 | 11
Vaginal hemorrhage (Reproductive system and breast disorders) | 8 | 5
Vaginal pain (Reproductive system and breast disorders) | 1 | 8
Vaginal stricture (Reproductive system and breast disorders) | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 10
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 14
Hot flashes (Vascular disorders) | 13 | 11
Hypertension (Vascular disorders) | 7 | 8

LIMITATIONS AND CAVEATS:
Some outcome measures were analyzed at a later time ("[later analysis]") and included a patient initially considered to be ineligible (protocol violation), but later deemed eligible, thus resulting in an additional participant for these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.